CLINICAL TRIAL: NCT02287883
Title: The Comparative Impact of Patient Activation and Engagement on Improving Patient-Centered Outcomes of Care in Accountable Care Organizations
Brief Title: Impact of Patient Activation and Engagement on Patient-Centered Outcomes of Care in ACOs
Acronym: ACTIVATE
Status: Completed | Type: Observational
Sponsor: University of California, Berkeley (Other)
Collaborators: Dartmouth College (Other); Wake Forest University Health Sciences (Other); HealthCare Partners Institute for Applied Research and Education (Unknown)
Responsible Party: Sponsor
Other Study IDs: IHS-1310-06821
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-10

CONDITIONS: Diabetes; Cardiovascular Disease
Keywords: Patient activation and engagement; Patient reported outcomes; Accountable Care Organizations; Chronic illness; Vulnerable population; Comparison of approaches
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Patient Participation; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients at high PAE clinic: Patients with diabetes or cardiovascular disease receiving care within two Accountable Care Organizations (ACOs) at clinics with high implementation of patient activation and engagement activities.
  Observational: Patient Activation and Engagement (PAE)
  Interventions: Other: Observational: Patient Activation and Engagement (PAE)
- Patients at low PAE clinic: Patients with diabetes or cardiovascular disease receiving care within two Accountable Care Organizations (ACOs) at clinics with low implementation of patient activation and engagement activities.
  Observational: Patient Activation and Engagement (PAE)
  Interventions: Other: Observational: Patient Activation and Engagement (PAE)

INTERVENTIONS:
Other: Observational: Patient Activation and Engagement (PAE) — Observational: Patients receive care from clinics with either low or high levels of patient activation and engagement activities.

SUMMARY:
The investigators will study the delivery of care to patients with diabetes and cardiovascular diseases from 16 practices in health care organizations who receive incentives for improving the quality of patient care. Half of those will be far along in engaging patients in their care and half will not. The investigators will see whether patients with diabetes or cardiovascular diseases who receive care from practices that more fully involve their patients have better clinical outcomes and satisfaction with their care than those who do not. The investigators expect that these findings will help practices and patients to achieve better outcomes of care.

DETAILED DESCRIPTION:
BACKGROUND Engaged patients have been referred to as "…the blockbuster drugs of the 21st century". Under the Affordable Care Act (ACA), Accountable Care Organizations (ACOs) are required to engage patients. The specific question we will address is: Do patients receiving care from ACO practices with highly developed patient activation and engagement (PA&E) activities achieve better patient reported health outcomes, report better experiences of care, and have better selected clinical measures (blood pressure, hemoglobin levels, and LDL-C) compared to patients receiving care from ACO practices with less developed PA&E initiatives? We plan to capitalize on the natural occurring variation in degree of implementing PA&E activities.

OBJECTIVES

1) To collect information on the PA&E activities in 16 practices of two ACOs at baseline and over three years - including initiatives focused on disease prevention and health promotion, care team-patient communication, shared decision-making, self-management support, advanced serious illness care, and patient involvement in the care redesign experience; 2) to assess the differences on patient-reported outcomes of care, patient experiences, and selected clinical measures between patients exposed to highly developed PA&E initiatives versus those receiving care from practices with minimal PA&E activities; and 3) examine practice-level variation in PA&E implementation processes including culture, leadership, teamwork, and relational coordination.

METHODS We will take advantage of the naturally occurring variation in the implementation of PA&E activities in 16 practices of two ACOs treating patients with diabetes and cardiovascular disease (CVD). A random sample of chronically-ill patients from each of the two ACOs will be sampled and will complete a patient-reported outcome instrument that includes select Patient-Reported Outcomes (PROMIS) measures and patient experience measures in early and late stages of the project. They will also complete the patient activation measure (PAM). We will examine changes over time in the outcome variables noted above. We will also survey ACO/ practice stakeholders regarding organizational culture, leadership, team effectiveness, and relational coordination using previously validated instruments supplemented by site visits. Multilevel analyses examine PA&E effects and practice-level heterogeneity within ACOs, controlling for patient characteristics.

PATIENT OUTCOMES The proposed project's explicit focus on examining the PA&E activities of ACO practices with highly developed PA&E activities in comparison with those with very little and linking these to the outcomes measures noted above should be of great interest to patients, the Patient-Centered Outcomes Research Institute (PCORI), and the health care policy and practitioner community. The findings should help to guide PCORI's future research agenda in this area while providing all involved with knowledge to advance patient-centered care.

ELIGIBILITY:
Inclusion Criteria:

* adult, 18-82
* diagnosis of diabetes or cardiovascular disease
* receives primary care at one of 16 selected clinical sites from two Accountable Care Organizations

Exclusion Criteria:

* Incomplete mailing address available from Electronic Medical Record
* Patient language other than English or Spanish

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4368 patients with diabetes or cardiovascular disease receiving care from selected clinics at two Accountable Care Organizations in Los Angeles, CA and Chicago, IL.
Sampling Method: Probability Sample
Enrollment: 2176 (Actual)
Dates: Start 2015-04; Primary Completion 2017-03 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Shortell, PhD,MPH,MBA, Principal Investigator — University of California, Berkeley
Locations (4):
- United States (4):
  - University of California, Berkeley, Berkeley, California
  - HealthCare Partners Insitute for Applied Research and Education, Torrance, California
  - Advocate Health Care, Chicago, Illinois
  - Dartmouth Colelge, Hanover, New Hampshire

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with diabetes and/or cardiovascular disease from sixteen primary care practice sites at two Accountable Care Organizations (ACOs) in the US (greater Los Angeles and Chicago areas) were surveyed about their patient reported outcomes (PROs), patient assessment of chronic illness care (PACIC) and patient activation and engagement (PAM).
Pre-assignment Details: Sixteen primary care practices at two ACOs in the US (greater Los Angeles and Chicago), were selected based on their responses to a 39-item questionnaire of their patient activation and engagement activities. 4168 eligible patients from these sites were included in the baseline survey. 2176 of these patients responded and were included in the study
Groups:
- Patients at High PAE Practices (n=8 Practices): Patients with diabetes or cardiovascular disease receiving care within two Accountable Care Organizations (ACOs) at practices with high implementation of patient activation and engagement (PAE) activities (top quartile).
- Patients at Low PAE Practices (n=8 Practices): Patients with diabetes or cardiovascular disease receiving care within two Accountable Care Organizations (ACOs) at practices with low implementation of patient activation and engagement (PAE) activities (bottom quartile).
Period: Overall Study
Arm/Group | Patients at High PAE Practices (n=8 Practices) | Patients at Low PAE Practices (n=8 Practices)
Started | 1081 | 1095
One-year Follow-up Survey | 622 | 669
Completed | 622 | 669
Not Completed | 459 | 426
Not completed — Death | 8 | 7
Not completed — No longer eligible | 222 | 182
Not completed — Non-response to survey | 229 | 237

BASELINE CHARACTERISTICS:
Groups:
- Patients at High PAE Practices: Patients with diabetes or cardiovascular disease receiving care within two Accountable Care Organizations (ACOs) at practices with high implementation of patient activation and engagement (PAE) activities.
- Patients at Low PAE Practices: Patients with diabetes or cardiovascular disease receiving care within two Accountable Care Organizations (ACOs) at practices with low implementation of patient activation and engagement (PAE) activities.
- Total: Total of all reporting groups
Arm/Group | Patients at High PAE Practices | Patients at Low PAE Practices | Total
Number analyzed (Participants) | 1081 | 1095 | 2176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 491 | 513 | 1004
  >=65 years | 590 | 582 | 1172
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 599 | 592 | 1191
  Male | 482 | 503 | 985
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 371 | 358 | 729
  Not Hispanic or Latino | 668 | 699 | 1367
  Unknown or Not Reported | 42 | 38 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 5 | 13
  Asian | 89 | 107 | 196
  Native Hawaiian or Other Pacific Islander | 4 | 5 | 9
  Black or African American | 230 | 35 | 265
  White | 412 | 601 | 1013
  More than one race | 22 | 27 | 49
  Unknown or Not Reported | 316 | 315 | 631
Patient Activation Measure (PAM-13) [Mean (Standard Deviation); unit: units on a scale] — Unweighted average of responses to 13-item Patient Activation Measure (PAM-13) which assesses patient knowledge, skill, and confidence for self-management. Response categories for all items range from 1 (disagree strongly with statements of activation) -4 (agree strongly with statements of activation).
  units on a scale | 3.27 (0.45) | 3.27 (0.44) | 3.27 (0.45)
Patient Assessment of Chronic Illness Care (PACIC) [Mean (Standard Deviation); unit: units on a scale] — Unweighted average of responses to 11-item Patient Assessment of Chronic Illness Care (PACIC). PACIC measures patients' experience with care they received from their health care providers with for their chronic condition. The response scale for all items ranges from 1 (never experienced care management process) -4 (always experienced care management process).
  units on a scale | 2.72 (0.83) | 2.65 (0.84) | 2.68 (0.83)
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form 8a [Mean (Standard Deviation); unit: units on a scale] — Patient Reported Social Functioning, scale 1 (never trouble or limited)-5 (always trouble or limited)
  units on a scale | 2.37 (1.03) | 2.34 (1.06) | 2.35 (1.05)
Patient Reported Outcomes Measurement Information System (PROMIS) Short Form 12a [Mean (Standard Deviation); unit: units on a scale] — Patient-Reported Physical Functioning, scale 1 (no difficulty) -5 (unable to do activity)
  units on a scale | 2.01 (0.89) | 1.99 (0.88) | 2.00 (0.88)
Patient Health Questionnaire 4 (PHQ-4) [Mean (Standard Deviation); unit: units on a scale] — Patient Reported Emotional Functioning, scale 1 (not at all anxious or depressed) -5 (anxious or depressed nearly every day)
  units on a scale | 1.55 (0.75) | 1.51 (0.72) | 1.53 (0.74)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 133.11 (14.99) | 130.31 (13.19) | 131.70 (14.18)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 76.14 (8.65) | 75.47 (8.10) | 75.80 (8.39)
Low density lipoprotein cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 91.82 (32.27) | 90.58 (31.50) | 91.22 (31.89)
Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage] | 7.33 (1.63) | 7.20 (1.49) | 7.27 (1.57)

OUTCOME MEASURES:

1. Primary Outcome: PROMIS Short Form 8a
Description: Patient Reported Social Functioning, scale 1 (always trouble or limited)-5 (never trouble or limited). Outcome measure is the mean of the change in scores reported by each patient between baseline (2015) and at one-year follow-up (2016).
Time Frame: 1 year
Population: Patients who completed surveys at both baseline (2015) and at one year follow-up (2016).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients at High PAE Practices | Patients at Low PAE Practices
Number analyzed (Participants) | 617 | 674
units on a scale | -0.05 (0.83) | -0.03 (0.86)
Statistical Analysis 1: Comparison: Patients at High PAE Practices vs Patients at Low PAE Practices; Test type: Other — Clustered two-sample t-test; p = 0.80, t-test, 2 sided

2. Primary Outcome: PROMIS Short Form 12a
Description: Patient-Reported Physical Functioning, scale 1 (unable to do activity) -5 (no difficulty). Outcome measure is the mean of the change in scores reported by each patient between baseline (2015) and at one-year follow-up (2016).
Time Frame: 1 year
Population: Patients completing a survey at both baseline (2015) and one-year follow-up (2016).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients at High PAE Practices | Patients at Low PAE Practices
Number analyzed (Participants) | 617 | 674
units on a scale | -0.07 (0.51) | -0.05 (0.55)
Statistical Analysis 1: Comparison: Patients at High PAE Practices vs Patients at Low PAE Practices; Test type: Other — Clustered two-sample t-test; p = 0.48, t-test, 2 sided

3. Primary Outcome: PHQ-4
Description: Patient Reported Emotional Functioning, scale 1 (anxious or depressed nearly every day) -5 (not at all anxious or depressed). Outcome measure is the mean of the change in scores reported by each patient between baseline (2015) and at one-year follow-up (2016).
Time Frame: 1 year
Population: Patients who completed a survey at both baseline and at one-year follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patients at High PAE Practices | Patients at Low PAE Practices
Number analyzed (Participants) | 617 | 674
units on a scale | 0.03 (0.62) | -0.04 (0.57)
Statistical Analysis 1: Comparison: Patients at High PAE Practices vs Patients at Low PAE Practices; Test type: Other — Clustered two-sample t-test; p = 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 3 years (January 2014-December 2016)
Description: We collected information annually on all-cause mortality occurring the prior calendar year. We did not collect other information about Serious Adverse Events or non-serious adverse events.
Arm/Group | Patients at High PAE Practices | Patients at Low PAE Practices
All-Cause Mortality (participants affected / at risk) | 14/1081 | 14/1095
Serious Adverse Events (participants affected / at risk) | 0/1081 | 0/1095
Other Adverse Events (participants affected / at risk) | 0/1081 | 0/1095

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-01-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT02287883/Prot_SAP_000.pdf
  • Informed Consent Form (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/83/NCT02287883/ICF_001.pdf